CLINICAL TRIAL: NCT06776874
Title: Studio Osservazionale Per lo Sviluppo di Uno Score Predittivo Degli Eventi Avversi Post-colangiopancreatografia Retrograda Endoscopica (ERCP)
Brief Title: Observational Study to Develop a Predictive Score for Adverse Events Post ERCP
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ADVERCP
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing ERCP according to normal clinical practice: The validation of the present predictive model and the one already published in the Literature will involve the simple application of the two models to a cohort of patients (so-called validation group), undergoing ERCP according to normal clinical practice; therefore, there will be no interventions that would may alter the patient's normal course of treatment.

SUMMARY:
The main objective of the study is: the identification of independent factors associated with an increased risk of post-ERCP complications. Other objectives are: the development of a predictive model of events post-ERCP adverse events and its validation; geographic validation of a predictive model already published in the literature using data collected during the study and the evaluation of the rate of post-ERCP AEs in the centers involved in the study.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) was described for the first time in 1968 and today is the pivotal procedure for the treatment of various biliopancreatic diseases. ERCP is associated with adverse events (AEs) such as post-ERCP pancreatitis (PEP), cholangitis and also with mortality.AEs related to therapeutic ERCP have been variably reported in several studies, with an estimated range of 4-30% for all AEs and 0.1-1% for overall mortality. In a systematic review of 21 studies prospective studies found an overall AE rate of 6.85% with mortality of 0.33%. PEP (3-15%) and bleeding (1-5%) are the two most common AEs, followed by cholangitis (1-5%) and perforation (1-2%). Several studies have attempted to identify potential risk factors for EAs ERCP-relati. Many of these studies are limited by the heterogeneity of definitions, the use of outdated criteria for the definition of AEs and by not large samples of patients. A more precise identification of the risk factors of EA related to ERCP is important so that preventive therapies can be introduced early and more effectively monitor individuals at increased risk. A recent retrospective study by Eduardo-Rodrigues Pinto et al. conducted on 1491 consecutive patients undergoing 1991 ERCP procedures, identified, based on pre- and intra-procedural covariables, risk factors related to patient and procedure for EA, in order to develop, through a multivariate logistic regression analysis, a predictive score estimating the likelihood of the occurrence of EA post-ERCP. This would allow a more correct information to the patient about the procedure and an optimization of the decision making of the physician in charge of the patient. Two two models, one considering only pre-procedural factors (model 1) and the other that considers both pre- and intra-procedural factors (model 2); both showed moderate predictive ability (AUC-ROC of 0.668 and 0.684 respectively). The score is based on data from patients from a single institution and has not been validated prospectively or externally to the population on which it was developed. The main objective of the study is: the identification of independent factors associated with an increased risk of post-ERCP complications. The secondary objectives are: the development of a predictive model of events post-ERCP adverse events and its validation; geographic validation of a predictive model already published in the literature [12] using data collected during the study and the evaluation of the rate of post-ERCP AEs in the centers involved in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients admitted with hepato-biliary-pancreatic disease or other pathological conditions that require treatment by ERCP
* Obtaining informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing ERCP according to normal clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 981 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
post-ERCP complications | 14 days
  Identification of independent factors associated with an increased risk of post-ERCP complications.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Lorenzo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No